CLINICAL TRIAL: NCT06559436
Title: Extending the Time Window for Intravenous Tenecteplase in Patients With Distal Medium Vessel Occlusions Stroke-a Randomised, Controlled, Multicentre Study
Brief Title: Extending the Time Window for Intravenous Tenecteplase in Patients With Distal Medium Vessel Occlusions Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of University of Science and Technology of China (Other)
Responsible Party: Principal Investigator, Wei Hu, Professor, The First Affiliated Hospital of University of Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNK-MeVO
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke
Keywords: Medium Vessel Occlusion; Stroke Due To Medium Vessel Occlusion; Beyond optimal time window; TNK intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous thrombolysis (Experimental): Patients in the TNK treatment group will receive TNK intravenous thrombolysis after MeVO is determined, and the usual dosage for TNK intravenous thrombolysis is 0.25mg/Kg, with a maximum of 25mg.
  Interventions: Drug: Intravenous thrombolysis
- Standard medical management (Active Comparator): Standard medical management
  Interventions: Other: Standard medical management

INTERVENTIONS:
Drug: Intravenous thrombolysis — Patients in the TNK treatment group will receive TNK intravenous thrombolysis after MeVO is determined, and the usual dosage for TNK intravenous thrombolysis is 0.25mg/Kg, with a maximum of 25mg,
  Arms: Intravenous thrombolysis
Other: Standard medical management — Standard medical management
  Arms: Standard medical management

SUMMARY:
To assess the safety and efficacy of beyond time window TNK intravenous thrombolysis for distal Medium Vessel Occlusion (MeVO) related stroke in a prospective randomized clinical trial.

DETAILED DESCRIPTION:
Previous study has confirmed that in acute ischemic stroke patients with large vessel occlusion within 4.5-24 hours of symptom onset and a salvageable penumbra on perfusion imaging, TNK thrombolysis is safe and can significantly improve the prognosis in the absence of mechanical thrombectomy. However, it is currently unknown whether TNK intravenous thrombolysis beyond optimal time window can improve the prognosis of distal Medium Vessel Occlusion (MeVO) related patients.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a primary (e.g., not secondary to endovascular therapy of proximal vessel occlusion) distal medium vascular occlusion defined as occlusion of the co/non-dominant M2 segment*, M3, or M4 segment of the middle cerebral artery (MCA), the anterior cerebral artery (ACA) (A1, A2, A3, or A4 segments), or the posterior cerebral artery (PCA) (P1, P2, P3, or P4 segments);

   * Co/non-dominant M2 segment vessel diameter should not exceed 2.0 mm. Co-dominant supplying 50% of the MCA territory vs non-dominant supplying <50% of the MCA territory.
2. Age ≥18 years;
3. Premorbid mRS 0-1;
4. Evidence of a disabling stroke defined as follows:

   1. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥4 at the time of randomization.
   2. NIHSS 2-3 with disabling deficit including significant aphasia, neglect, hemianopsia, or hemiparesis/ loss of hand or leg function as established by the treating team in context of the patient's life.
5. Less than 50% core in the territory supplied by the occluded vessel as evident by hypodensity and loss of grey-white border on NCCT or ADC <620 mm2/s on diffusion MRI or rCBF<30% on CTP after 6h of symptom onset.
6. Time from onset (or time last seen well) to treatment within 4.5-24 hours;
7. Informed consent obtained from patient or acceptable patient surrogate.

Exclusion Criteria:

1. Received intravenous thrombolysis prior to randomization;
2. Allergy to Tenecteplase;
3. Seizures, or other neurological/mental illness at stroke onset if it precludes obtaining an accurate baseline NIHSS;
4. Patients planned to undergo MT or other endovascular treatments (e.g., intra-arterial thrombolysis);
5. Systolic blood pressure>185 mmHg or diastolic blood pressure>110 mmHg, which cannot be controlled by antihypertensive drug(s);
6. Acute intracerebral hemorrhage identified by CT or MRI;
7. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal;
8. Subjects with occlusions in multiple vascular territories (e.g., bilateral or multi-territorial anterior circulation, or anterior/posterior circulation);
9. Contraindication to imaging with MR or CT with contrast agents;
10. Known genetic or acquired bleeding diathesis, or received warfarin and INR > 1.7; or treated with direct oral anticoagulant agents in the prior 48 hours;
11. Platelets <100×109/L, APTT > 40 s, or PT >15 s; Blood glucose <50 mg/dl (2.7 mmol/L) or >400 mg/dl (22.2 mmol/L);
12. Severe renal failure, defined as serum creatinine > 3.0 mg/dl (or 265.2 μmol/l) or glomerular filtration rate (GFR) < 30, or patients requiring hemodialysis or peritoneal dialysis;
13. Active internal hemorrhage or at high risk of bleeding, e.g., major surgery, sever trauma or gastrointestinal or urinary tract hemorrhage within the last 2 weeks, or arterial puncture at a non-compressible site within the previous 7 days;
14. Ischemic stroke or myocardial infarction in previous 3 months, previous intracranial hemorrhage, severe traumatic brain injury or intracranial or intraspinal operation in previous 3 months, or known intracranial neoplasm, arteriovenous malformation or giant aneurysm;
15. Life expectancy < 1 year;
16. Patients who cannot adhere to the trial protocol or follow-up;
17. Currently participating in other clinical trials;
18. Pregnant or lactating women;
19. Any other condition that, in the opinion of the investigator, could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Rates of 90 day good functional outcomes | 90 (± 14 days) after procedure
  (mRS score ≤ 1 is defined as good prognosis)

SECONDARY OUTCOMES:
2. Proportion of patients with functional independence outcome (mRS 0-2) at day 90 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
3. Proportion of patients with ambulatory and self-care capable outcome (mRS 0-3) at day 90 | 90 (± 14 days) after procedure
  modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

OTHER OUTCOMES:
Symptomatic intracranial hemorrhage (sICH) | 24 hours after procedure
  SICH means any hemorrhage with neurological deterioration, as indicated by an NIHSS score that was higher by ≥4 points than the value at baseline or the lowest value in the first 24 hours , or any hemorrhage leading to death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No